CLINICAL TRIAL: NCT00327782
Title: Palliative Care of Children With End-Stage Heart Failure
Status: Terminated | Type: Observational
Sponsor: Children's Healthcare of Atlanta (Other)
Other Study IDs: 06-114
Record Dates: First submitted 2006-05-18; First posted 2006-05-19 (Estimated); Last update posted 2007-05-04 (Estimated); Status verified 2007-05

CONDITIONS: Congenital Disorders
Keywords: pediatric; palliative care; end stage heart failure
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Retrospective

SUMMARY:
Palliative care in pediatric oncology and neurology is well described in the literature. There is a lack of information on the care of children terminally ill due to heart failure. A significant number of children are diagnosed with terminal heart failure for which palliative care is required.

Objective:

To describe palliative care of children over one year of age with end-stage heart failure, including need for and types of pain control, hospice use, need for and use of home nursing and quality of life issues.

DETAILED DESCRIPTION:
Methods:

Retrospective chart review of all children over one year of age diagnosed with end-stage heart failure between January 1, 1995 and December 31, 2005 at Children's Healthcare of Atlanta, Egleston Hospital, followed by Sibley Heart Center Cardiology.

Patient variables taken from the medical charts will include:

Diagnosis Age, gender Medications Prior surgery or transplantation Associated conditions such as muscular dystrophy, renal failure

Practice variables taken from the medical charts will include:

Hospice care provided Home inotropic infusions Medications administered for pain Social work/psychology evaluation DNR status

Statistics:

Number of patients receiving home nursing, involved in hospice, treated with pain medications, home oxygen or home inotropes.

ELIGIBILITY:
Inclusion Criteria:

* Any patient between 1 - 18 years of age (inclusive) Any patient with end stage heart disease Treated at Egleston Hospital, Children's Healthcare of Atlanta Followed by Sibley Heart Center Cardiology

Exclusion Criteria:

* Those who do not meet inclusion criteria

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 1995-01; Study Completion 2006-04

CONTACTS AND LOCATIONS:
Overall Officials: William T Mahle, MD, Principal Investigator — Emory University SOM, Children's Healthcare of Atlanta
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States